CLINICAL TRIAL: NCT00966095
Title: A Prospective, Multi-Center PRostate Cancer Individual Signature Evaluation Trial (PReCISE) in Patients Undergoing Scheduled Prostate Biopsy
Brief Title: PRostate Cancer Individual Signature Evaluation Trial in Patients Undergoing Scheduled Prostate Biopsy
Acronym: PReCISE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Source MDx (Industry)
Responsible Party: Lisa Siconolfi, PhD, Director of Clinical Studies, Source MDx
Other Study IDs: PReCISE
Record Dates: First submitted 2009-08-24; First posted 2009-08-26 (Estimated); Last update posted 2010-11-25 (Estimated); Status verified 2010-11

CONDITIONS: Prostate Cancer
Keywords: prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood for gene expression analysis
  serum
  plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- men scheduled for prostate biopsy

SUMMARY:
The purpose of this study is to develop and validate a blood-based diagnostic test that will predict prostate biopsy outcome as positive or negative for prostate cancer. Such a test will serve to reduce the number of unnecessary prostate biopsies.

ELIGIBILITY:
Inclusion Criteria:.

1. Male over the age of 40.
2. Patient is scheduled for prostate biopsy for one or more of the following reasons:

   * PSA > 2.5 ng/ml
   * Rising PSA (>0.5 ng/ml/yr)
   * Lower PSA value with other risk factors for prostate cancer (e.g.; family history)
   * Abnormal DRE
   * Percent free PSA <15%
3. No prior history of prostate cancer or prostate biopsy.

Exclusion Criteria:

* Unable or unwilling to provide informed consent

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men scheduled for a prostate biopsy
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2009-12

PRIMARY OUTCOMES:
ability of whole blood gene expression to predict biopsy outcome | pre-biopsy

SECONDARY OUTCOMES:
Prediction of tumor aggressiveness using whole blood gene expression | post-biopsy

CONTACTS AND LOCATIONS:
Overall Officials: William Oh, MD, Principal Investigator — Mt. Sinai School of Medicine; Danute "Bunki" Bankaitis-Davis, PhD, Principal Investigator — Source MDx; Lisa Siconolfi, PhD, Principal Investigator — Source MDx; Philip Kantoff, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (17):
- United States (17):
  - San Bernardino Urological Associates, San Bernardino, California
  - The Urology Center of Colorado, Denver, Colorado
  - University of Chicago Medical Center, Chicago, Illinois
  - Johns Hopkins University Brady Urological Institute, Baltimore, Maryland
  - Brigham and Women's Hospital/ Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Bay State Clinical Trials, Watertown, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Karmanos Cancer Institute Wayne State University, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University Urology Associates, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Durham VA Medical Center, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Urology Clinics of North Texas, Dallas, Texas
  - Urology San Antonio Research, San Antonio, Texas
  - University of Washington Department of Urology, Seattle, Washington